CLINICAL TRIAL: NCT04642885
Title: Families Coping Together With Alzheimer's Disease
Acronym: FACT-AD
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2000024219; R01AG058565 (NIH)
Record Dates: First submitted 2020-11-20; First posted 2020-11-24 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Family Research; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dyad: parent with dementia and an adult child who is a caregiver

SUMMARY:
Two remote phone/zoom calls are required to assess experiences as a family coping with dementia.

DETAILED DESCRIPTION:
Using a combination of paper or online surveys in addition to interactive visits with blood pressure monitoring, participants are observed interacting with each other. Blood pressure devices are mailed to their homes and only worn for six minute intervals. The first visit generally lasts one hour and the second visit 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Parent must be 55 plus with symptoms or a diagnosis of dementia
* Adult child must be over 18 and involved in some way with assisting parent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, adult children of a parent over 55 with early stage dementia who are responsible for helping parent with at least one task will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Caregiver demand appraisals | Baseline and one year
  (1a) Caregiver demand appraisals: 6 items from the 12-item Zarit Burden Interview (ZBI) will assess caregiver appraisals of demands (e.g., That because of the time you spend with your relative that you don't have enough time for yourself?". Caregivers self-report aspects of burden on a scale from 0 (never) to 4 (nearly always; α= .86). Higher numbers indicate higher demands. Administration is 2.5 minutes
Caregiver perceived stress | Baseline and one year later
  (1b) Caregiver perceived stress: 6 items from the 12-item Zarit Burden Interview (ZBI) will assess caregiver perceived stress (e.g., "Stressed between caring for your relative and trying to meet other responsibilities (work/family)?"). Caregivers self-report aspects of burden on a scale from 0 (never) to 4 (nearly always; α= .86). Higher numbers indicate higher stress. Administration is 2.5 minutes.
Caregiver negative Coping | Baseline and one year later
  The Brief COPE Inventory is a shortened version (28 items) of the COPE inventory in which respondents indicate how often they use a particular coping strategy under stress as ranked on a 4-point scale with 1 (I haven't been doing this at all) to 4 (I've been doing this a lot). Examples of items include "I've been using alcohol or drugs to help me get through it." and "I've been criticizing myself" (α=0.72, 0.84, 0.75 for emotion, problem, and dysfunction focused subscales). Higher scores indicate poorer coping. Administration is 10 minutes

SECONDARY OUTCOMES:
Relational Functioning | Baseline and one year later
  The Relationships Inventory will measure the degree to which individuals perceive that they can rely on their parent or child for help and support when needed (e.g., "to what extent can you count on your parent/child for help with a problem?" "to what extent can you count on your parent/child to give you honest feedback, even when you might not want to hear it?"). Ratings will be made on a scale from 1 (not at all) to 5 (very much; α=.79). Four additional items will assess the degree to which individuals perceive that their parent/child is a good support-provider (e.g., "overall, my parent/child is a good support-provider" using a scale from 1 (strongly disagree) to 7 (strongly agree). Higher numbers indicate higher relationship functioning. Administration is 5 minutes.
Health | Baseline and one year later
  Health-related quality of life will be assessed using the 12-item Short Form Survey (SF-12) version 1.0, documenting the extent of limitations in a number of domains. Higher scores indicate better physical and mental health-related quality of life. It has been used with both persons with ADRD and caregivers. Administration is 5 minutes. The minimum and maximum scores are 0 and 100.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Monin, PhD, Principal Investigator — Yale University
Locations (1):
- Yale school of Public Health, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT04642885/ICF_000.pdf